CLINICAL TRIAL: NCT03986827
Title: A Disorder Specific Group Cognitive Behavior Therapy for Social Anxiety Disorder in Adolescents
Brief Title: Cognitive Behavioral Therapy for Adolescents With Social Anxiety Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Aarhus (Other)
Collaborators: TRYG Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 124958; 124958 (Other Grant/Funding Number: TRYG Foundation)
Record Dates: First submitted 2019-06-06; First posted 2019-06-14 (Actual); Last update posted 2019-06-24 (Actual); Status verified 2019-04

CONDITIONS: Social Anxiety Disorder
Keywords: Social anxiety disorder; Social phobia; Youth; Cognitive behavioral therapy; Adolescents
MeSH Terms: conditions — Phobia, Social

STUDY DESIGN:
Intervention Model Description: The study is a randomized controlled superiority trial comparing two active groups of treatment: 1) Cool Kids Anxiety Program - Social Enhanced (CK-E), 2) Cool Kids Anxiety Program (CK). The study design is a mixed between-within design, with data points pre- and post-treatment, and at 3- and 12-month follow-ups.
Who Masked: Participant, Outcomes Assessor
Masking Description: Randomization will be stratified into two age groups (12-14 and 15-17) using permuted block design with a fixed block size of 8 at a 1:1 ratio to the CK or the CK-E condition. Randomization will be conducted with an online computer random number generator (www.random.org) by an independent secretary. The sequence list will be kept concealed from therapists until treatment starts. Participants are not informed about their specific treatment condition.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cool Kids Anxiety Program - Social Enhanced (CK-E) (Experimental): CK-E is a G-CBT treatment developed specifically for treatment of youth SAD. The program consists of 10 2-h group sessions with four to five adolescents and their parents in each group. 9 sessions with the adolescents and parents together and one parents-only session (session 5). Three months after ending treatment participant will be offered a 1-h booster group session.
  Interventions: Behavioral: Cool Kids Anxiety Program - Social Enhanced
- Cool Kids Anxiety Program (CK) (Active Comparator): The standard Cool Kids Anxiety Program is a treatment program based on generic CBT techniques such as cognitive restructuring and gradual exposure.
  The program consists of 10 2-h group sessions with four to five adolescents and their parents in each group. 9 sessions with the adolescents and parents together and one parents-only session (session 5). Three months after ending treatment participant will be offered a 1-h booster group session.
  Interventions: Behavioral: Cool Kids Anxiety Program

INTERVENTIONS:
Behavioral: Cool Kids Anxiety Program - Social Enhanced — Specific G-CBT intervention for adolescents with social anxiety disorder
  Other Names: CK-E
  Arms: Cool Kids Anxiety Program - Social Enhanced (CK-E)
Behavioral: Cool Kids Anxiety Program — Generic G-CBT intervention for adolescents with anxiety disorders
  Other Names: CK
  Arms: Cool Kids Anxiety Program (CK)

SUMMARY:
The main aim of the present study is to investigate the effectiveness of a disorder specific group cognitive behavior therapy (G-CBT) program for youth SAD, the, Cool Kids Anxiety Program - Social Enhanced (CK-E), developed at Macquarie University, Sidney, Australia.

Furthermore, the study will examine how well this program fares against generic CBT treatment.

DETAILED DESCRIPTION:
The main aim of the study is to investigate the effectiveness of a disorder specific G-CBT program for youth SAD compared to a generic G-CBT program for anxiety disorders.

Reduction in anxiety symptoms is expected for both treatment conditions although we hypothesize better outcome for the enhanced treatment condition.

Approximately 96 adolescents aged 12 to 17 years will be included with data points at pre- and post-treatment, and at 3-month and 1-year follow-ups.

ELIGIBILITY:
Inclusion Criteria:

* Youth between 12 and 17 years of age.
* Social anxiety disorder as the primary disorder measured using the Anxiety Disorder Interview Schedule for DSM-IV, Child and Parent Version (ADIS-IV C/P).

Exclusion Criteria:

* A diagnosed autism spectrum disorder (ASD).
* Untreated Attention Deficit Hyperactivity Disorder (ADHD).
* Psychotic symptoms.
* Current severe self-harm or suicidal ideation.
* Current eating disorder.
* CSR>5 on depression.
* Received prior CK treatment within the last two years.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 96 (Estimated)
Dates: Start 2019-02-28 (Actual); Primary Completion 2022-02-28 (Estimated); Study Completion 2022-05-28 (Estimated)

PRIMARY OUTCOMES:
Change in social anxiety disorder symptoms - measured using Anxiety Disorder Interview Schedule for DSM-IV, Child and Parent Version (ADIS-IV C/P) | Baseline, post-treatment (after session 10 = 10-14 weeks after baseline interview) and follow-up 3-month after session 10.
  ADIS-IV C/P is a semi-structured diagnostic interview conducted with youth and parents separately to assess the diagnostic criteria for anxiety disorders in accordance with DSM-IV as well as other disorders often comorbid with anxiety (e.g., depression and ADHD). Severity of the diagnosis is measured on a nine-point Likert scale ranging from not disturb at all to severely disturbed (0-8). CSR scores of 4 or greater indicate a clinical diagnosis. Separate CSRs are made by youths, parents, and the clinician, but only the CSRs provided by the clinician will be used. The most impairing diagnosis, as assessed by the clinician, will be considered as the primary diagnosis.
Change in social anxiety disorder symptoms - measured using The Social Phobia Inventory (SPIN) | Baseline, post-treatment (after session 10 = 10-14 weeks after baseline interview) and follow-ups at 3- month and 1-year after session 10.
  The Social Phobia Inventory (SPIN) (Connor et al., 2000). SPIN is a questionnaire used for measuring youths self-rated SAD symptoms. It includes 17 items covering SAD symptoms of fear, avoidance and physiological/bodily reactions (trembling, blushing, heart palpitations and sweating). The adolescents are asked to which degree they have been bothered by these symptoms the preceding week. Each item is rated on a five-point Likert scale (0-4). Higher scores indicate higher degree of distress regarding the symptom. The SPIN has been found to have good internal consistency, test-retest reliability, and convergent and divergent validity (M. M. Antony, Coons, McCabe, Ashbaugh, & Swinson, 2006; Connor et al., 2000). The SPIN has demonstrated good psychometric properties for assessing youth SAD (Ranta, Kaltiala-Heino, Koivisto, et al., 2007; Ranta, Kaltiala-Heino, Rantanen, Tuomisto, & Marttunen, 2007; Tsai, Wang, Juang, & Fuh, 2009)
Change in social anxiety disorder symptoms - measured using Spence Children's Anxiety Scale (SCAS and SCAS-P) | Baseline, post-treatment (10-14 weeks), 3-month follow-up and 1-year follow-up
  is used to measure adolescent- and parent-rated anxiety symptoms. The adolescent version contains 44 items (including six positive filler items), and the parent version contains 38 items. Items are rated on a four-point Likert scale (0-3). Higher scores indicate higher levels of anxiety. It consists of six subscales reflecting symptoms specifically related to social phobia, panic disorder and agoraphobia, generalized anxiety disorder, obsessive-compulsive disorder, separation anxiety disorder, and fear of physical injury

SECONDARY OUTCOMES:
The Child Anxiety Life Inference Scale (CALIS) | Baseline, post-treatment (10-14 weeks), 3-month follow-up and 1-year follow-up
  is used to measure the impact of youth's anxiety on various areas of life functioning including friends, school, extracurricular, and family. The impact is evaluated separately by adolescents (9 items) and their parents (16 items). Items are evaluated on a five point Likert scale (0-4). Higher scores indicate a higher degree of life interference.
The Short version of the Mood and Feelings Questionnaire (S-MFQ) | Baseline, post-treatment (10-14 weeks), and 3-month follow-up
  will be used in the present study to measure depressive symptoms within the last two weeks. The symptoms are evaluated independently by adolescents and parents. The short version includes 13 items rated on a three-point Likert scale.
The Negative Effects Questionnaire (NEQ) | posttreatment (10-14 weeks)
  dis a self-administered measure of negative effects of psychological treatment. For this specific study we adjusted the NEQ for the age group (12-17) and their parents. Both adolescents and parents are to complete the NEQ. NEQ consists of three parts. First, participants endorse whether a specific item has occurred during treatment (yes/no). Secondly, participants rate how negatively the effect was on a 4-point Likert scale, ranging from "not at all" to "extremely" (0-4). Third, they attribute the negative effect to either "the treatment they receive" (1) or "other circumstances" (0).
The Child Health Utility 9D (CHU 9D) | posttreatment (10-14 weeks)
  is developed to determine how health affects children's lives. In this study CHU 9D is rated by the adolescents. CHU 9D is a generic preference-based self-rated measurement of health-related quality of life. It consists of nine dimensions; worry, sadness, tiredness, pain, annoyed feeling, school work, daily routine, sleep, and activities. These nine dimensions each have five levels on which the adolescents rates the level to how they are feeling.

OTHER OUTCOMES:
Background information | Baseline, post-treatment (10-14 weeks), 3-month follow-up and 1-year follow-up
  Parents will complete a background questionnaire pretreatment. This questionnaire includes information regarding parents' mental and physical health, adolescent's mental and physical health, family demographics, household income and parents level of education, adolescent's previous and/or ongoing treatment, school absenteeism, and developmental point of orientation.
Credibility/expectation questionnaire (CEQ ) | CEQ will be completed after session 1 (week one)
  is a self-rated measure addressing the participants' expectancy and credibility of the treatment. Both youth and parents complete the questionnaire. CEQ consists of 6 items; three items regarding credibility and three items regarding expectancy.
Experience of Service Questionnaire (ESQ) | posttreatment (10-14 weeks)
  measures participants' satisfaction with the intervention. ESQ is adjusted by CEBU from the Experience of Service Questionnaire (Attride-Stirling, 2002). There are separate items for parents (10 items) and adolescents (7 items). ESQ includes both positive and negative statements, and items are rated on a 3-point Likert scale.
Depression Anxiety Stress Scales (DASS) | Baseline, post-treatment (10-14 weeks), 3-month follow-up
  is used in the study for parents' rating of their own symptoms regarding anxiety, depression and stress. DASS consists of three subscales measuring symptoms of anxiety (DASS-A), depression (DASS-D) and stress (DASS-S). DASS contains 42 item and each item is rated on a four-point Likert scale (0-3) with higher scores indicating a higher degree of distress.
Mini-SPIN | In the current study mini-SPIN will be used as a severity measure rated by the adolescents prior to session 1 (week one), 4 (week four), 7 (week seven) and 10 (week 10-14)
  is developed as a brief screening instrument for SAD but can also serve as a repeated outcome measurement. The mini-SPIN is completed by the adolescents themselves. Mini-SPIN includes three specific items from the original SPIN ("Fear of embarrassment causes me to avoid doing things or speaking to people"; "I avoid activities in which I am the center of attention"; and "Being embarrassed or looking stupid is among my worst fears"). Each item is rated on a five-point Likert scale (0-4).
Postevent version of the Thoughts Questionnaire (PTQ) | Assessed after session session 1 (week one), 4 (week four), 7 (week seven) and 10 (week 10-14)
  is self-rated measure to assess the degree of post event processing. Adolescents complete the PTQ. Consistent with prior research (Perini, Abbott, & Rapee, 2006; Wong et al., 2017) only the 15 negatively worded items of the PTQ will be used in this study.
Focus of Attention Questionnaire (FAQ) | Adolescents complete FAQ after session session 1 (week one), 4 (week four), 7 (week seven) and 10 (week 10-14)
  is a self-rated measure of focus of attention. It is completed by the adolescents themselves. FAQ is a 10-item scale including two 5-item subscales; self-focused attention and external-focused attention. All items are rated on a five-point Likert scale ranging from 1-5 (1 = "Not at all", 5 = "Totally"). The two subscales are treated as independent.
Subtle Avoidance Frequency Examination (SAFE) | Baseline, post-treatment (10-14 weeks), 3-month follow-up
  is a self-rated measure designed to assess safety behaviors. In the study adolescents complete the questionnaire. SAFE is designed to incorporate both active safety behaviors, subtle restriction of behavior, and behaviors aimed at avoiding or concealing physical symptoms. SAFE consists of 32 items ranging on a five point Likert scale (0-4), with higher scores indicating a higher degree of safety-seeking behaviors.
The Children's Automatic Thoughts Scale (CATS) | Baseline, post-treatment (10-14 weeks), 3-month follow-up
  measures a range of the adolescents' self-reported negative self-statements. CATS is completed by the adolescents themselves. CATS include four subscales relating to automatic thoughts on social threat, personal failure, hostility, and physical threat. All items are scored on a five-point Likert scale (0-4), with higher scores indicating higher degrees of negative automatic thought. Only two subscales are included in the questionnaire battery of the present study; social threat and personal failure.

CONTACTS AND LOCATIONS:
Overall Officials: Mikael Thastum, Professor, Principal Investigator — University of Aarhus
Locations (1):
- Aarhus University, Department of Psychology and Behavioural Sciences, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Agersnap TN, Lomholt JJ, Jensen MB, Thastum M. Comparison of Disorder-Specific Group CBT and Generic Group CBT in Treating Adolescents with Social Anxiety Disorder: A Randomized Controlled Trial. Res Child Adolesc Psychopathol. 2026 Feb 6;54(1):27. doi: 10.1007/s10802-025-01412-z. PMID 41652081
- [Derived] Lassen NF, Hougaard E, Arendt KB, Thastum M. A disorder-specific group cognitive behavior therapy for social anxiety disorder in adolescents: study protocol for a randomized controlled study. Trials. 2019 Dec 21;20(1):757. doi: 10.1186/s13063-019-3885-3. PMID 31864383